CLINICAL TRIAL: NCT01159990
Title: A Randomized, Double Blind Phase 1b Trial to Examine the Influence of Antigenic Competition on the Immunogenicity of HIV-1 Gag/Pol: A Comparison of rAd5 Gag/Pol Env A/B/C to rAd5 Gag/Pol
Brief Title: Antigenic Competition in HIV Preventive Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 084; 10785 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombinant adenovirus serotype 5 (rAd5) Gag/Pol Env A/B/C (Experimental): Participants will receive one intramuscular injection of rAd5 Gag/Pol Env A/B/C.
  Interventions: Biological: rAd5 Gag-Pol Env A/B/C
- rAd5 gag/pol (Active Comparator): Participants will receive one intramuscular injection of rAd5 gag/pol.
  Interventions: Biological: rAd5 Gag-Pol

INTERVENTIONS:
Biological: rAd5 Gag-Pol Env A/B/C — 1×10^10 particle units (PU) rAd5 Gag-Pol, Env A/B/C (3:1:1:1 mixture) delivered via intramuscular injection
  Arms: Recombinant adenovirus serotype 5 (rAd5) Gag/Pol Env A/B/C
Biological: rAd5 Gag-Pol — 5×10^9 PU rAd5 Gag-Pol delivered via intramuscular injection
  Arms: rAd5 gag/pol

SUMMARY:
HIV vaccines are designed to create an immune response to certain components of the HIV virus called peptides. Previous research indicates that one peptide, called Gag, may be particularly important for stimulating an immune response to HIV. Many vaccines being studied combine multiple peptides, but including other peptides may weaken the body's response to Gag. This study will test whether a vaccine that targets Gag and another peptide called Env is better than a vaccine without Env at causing an immune response to Gag.

DETAILED DESCRIPTION:
HIV vaccines are designed to create an immune response to certain parts of the HIV virus called peptides. Researchers believe that eliciting a response to a peptide called Gag is particularly important. Most HIV vaccines in current clinical trials combine multiple peptides, but including these other peptides may cause antigenic competition. Antigenic competition occurs when the body's immune system reaction to one part of a vaccine weakens or inhibits the response to another part of the vaccine. Specifically, this study is concerned that having too many other peptides in a vaccine might weaken the specific immune response to Gag. This study will test whether a vaccine which only includes the peptides Gag and Pol elicits a stronger immune response to Gag and Pol than a vaccine that also includes the peptides Env A, B, and C.

Participation in this study will last 6 months. The number of study visits will vary by study site. Participants will be randomly assigned to receive injections of one of two vaccines in their upper arm. One group of participants will receive rAd5 gag/pol, which contains only the Gag and Pol peptides, while the other group of participants will receive rAd5 gag/pol Env A/B/C, which contains the Gag, Pol, and Env A, B, and C peptides. For 3 days after injection, participants will need to record their temperature and any side effects, and they will be contacted by study staff 7 days after the injection for follow-up monitoring.

During study visits, participants will complete the following assessments: an HIV test; a physical exam; collection of blood samples; a pregnancy test; and an interview about health, medications, HIV risk behaviors, and experiences with the study.

Participants will be contacted by study staff once a year for 5 years after the vaccination for follow-up health and safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HIV Vaccine Trials Network (HVTN) Clinical Research Site (CRS) and willingness to be followed for the planned duration of the study
* Completes a questionnaire prior to vaccination that demonstrates an understanding of this study and that in a previous trial there was an association of increased HIV acquisition with receipt of that study vaccine
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Willingness to continue annual follow-up contact after the last required protocol clinic visit, for a total of 5 years following enrollment
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Assessed by the clinic staff as being at low risk for HIV infection on the basis of sexual behaviors within the 12 months prior to enrollment
* Adenovirus 5 (Ad5) neutralizing antibody (nAb) titer less than 1:18
* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, or greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell (WBC) count between 3,300 and 12,000 cells/mm3
* Total lymphocyte count greater than or equal to 800 cells/mm3
* Remaining differential either within institutional normal range or with site physician approval
* Platelet count between 125,000 and 550,000/mm3
* Alanine aminotransferase (ALT) less than or equal to 1.25 times institutional upper limits of normal
* Negative HIV-1 and HIV-2 blood test: U.S. participants must have negative FDA-approved enzyme immunoassay (EIA). Non-U.S. sites may use locally available assays that have been approved by HVTN laboratory operations.
* Negative for Hepatitis B surface antigen (HBsAg)
* Negative for anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) test if the anti-HCV is positive
* Negative pregnancy test for female participants prior to vaccination on the day of vaccination
* Agreement to avoid pregnancy for female participants, either through abstinence or appropriate use of contraceptives
* If born male, must be fully circumcised (as documented at screening examination)

Exclusion Criteria:

* Within the 12 months prior to enrollment: excessive daily alcohol use, frequent binge drinking, chronic marijuana abuse, or any other use of illicit drugs
* Within the 12 months prior to enrollment: a history of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), Chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B virus
* Received non-HIV experimental vaccine(s) within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For potential participants who have received the control or placebo in an experimental vaccine trial, the HVTN 084 PSRT will determine eligibility on a case-by-case basis.
* For potential participants who received the control or placebo in an HIV vaccine trial, documentation of the identity of the study control or placebo must be provided to the HVTN 084 protocol safety review team (PSRT), who will determine eligibility on a case-by-case basis.
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, or abdominal pain. A participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child will not be excluded.
* Immunosuppressive medications received within 168 days before first vaccination, except (1) corticosteroid nasal spray for allergic rhinitis, (2) topical corticosteroids for mild, uncomplicated dermatitis, or (3) oral or parenteral corticosteroids given for non-chronic conditions not expected to recur (length of therapy 10 days or less with completion at least 30 days prior to enrollment).
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 60 days before first vaccination
* Live attenuated vaccines other than influenza vaccine received within 30 days before vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccines or any vaccines that are not live attenuated vaccines (e.g., tetanus, pneumococcal, hepatitis A or B), or allergy treatment with antigen injections that were received within 14 days prior to the vaccination
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the study
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, physical examination findings, abnormal laboratory results, or past medical history with implications for current health.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Angioedema (hereditary, acquired, or idiopathic) or idiopathic urticaria within the last 3 years if episodes are considered serious or have required medication within the last 2 years
* Autoimmune disease
* Immunodeficiency
* Untreated or incompletely treated syphilis infection
* Asthma other than mild, well-controlled asthma
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. History of isolated gestational diabetes does not mandate exclusion.
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Body mass index (BMI) greater than or equal to 40
* Hypertension that is not well controlled
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy. Not excluded: a participant with a surgical excision and subsequent observation period that, in the investigator's estimation, has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study.
* Seizure disorder. Not excluded: a participant with a history of seizures who has not required medications or had a seizure within the past 3 years.
* Asplenia, defined as any condition resulting in the absence of a functional spleen
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, persons at ongoing risk for suicide, or persons with a history of suicide attempt or gesture within the past 3 years.
* Pregnant or breastfeeding
* Has been fully circumcised within 90 days prior to first vaccination or displays evidence that surgical site is not fully healed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Magnitude of Gag and/or Pol-specific T-cell responses, as measured by Enzyme-Linked Immunospot (ELISpot) | Measured 4 weeks after immunization
Number of Gag and/or Pol epitopes targeted by CD4+ and CD8+ T-cells, as measured by ELISpot | Measured 4 weeks after immunization

SECONDARY OUTCOMES:
Number of individuals mounting T-cell responses to Gag and/or Pol, as assessed by ELISpot | Measured 4 weeks after immunization
Local and systemic reactogenicity signs and symptoms, laboratory measures of safety, adverse events (AEs), and AEs reported on an expedited basis to Division of AIDS (DAIDS) | Measured over 6 months after immunization
Magnitude of Gag and/or Pol-specific CD4+ and CD8+ T-cell responses, as measured by intracellular cytokine staining (ICS) | Measured 4 weeks after immunization

CONTACTS AND LOCATIONS:
Overall Officials: Esper Kallas, MD, PhD, Study Chair — University of Sao Paulo
Locations (7):
- United States (3):
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
- Sao Paulo HVTU - CRT DST/AIDS CRS, São Paulo, Brazil
- Peru (2):
  - ACSA CRS, Iquitos, Maynas
  - Barranco CRS, Lima
- Lausanne Vaccine and Immunotherapy Center CRS, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] McElrath MJ, De Rosa SC, Moodie Z, Dubey S, Kierstead L, Janes H, Defawe OD, Carter DK, Hural J, Akondy R, Buchbinder SP, Robertson MN, Mehrotra DV, Self SG, Corey L, Shiver JW, Casimiro DR; Step Study Protocol Team. HIV-1 vaccine-induced immunity in the test-of-concept Step Study: a case-cohort analysis. Lancet. 2008 Nov 29;372(9653):1894-1905. doi: 10.1016/S0140-6736(08)61592-5. Epub 2008 Nov 13. PMID 19012957
- [Background] Kiepiela P, Ngumbela K, Thobakgale C, Ramduth D, Honeyborne I, Moodley E, Reddy S, de Pierres C, Mncube Z, Mkhwanazi N, Bishop K, van der Stok M, Nair K, Khan N, Crawford H, Payne R, Leslie A, Prado J, Prendergast A, Frater J, McCarthy N, Brander C, Learn GH, Nickle D, Rousseau C, Coovadia H, Mullins JI, Heckerman D, Walker BD, Goulder P. CD8+ T-cell responses to different HIV proteins have discordant associations with viral load. Nat Med. 2007 Jan;13(1):46-53. doi: 10.1038/nm1520. Epub 2006 Dec 17. PMID 17173051